CLINICAL TRIAL: NCT01999608
Title: Vitamin D Deficiency and Ovarian Reserve Among Infertile Patients. A Cross-sectional Analysis
Brief Title: Vitamin D Deficiency and Ovarian Reserve Among Infertile Patients
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Nikolaos P. Polyzos, Principal Investigator, Universitair Ziekenhuis Brussel
Other Study IDs: 2013/180
Record Dates: First submitted 2013-11-18; First posted 2013-12-03 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-06

CONDITIONS: Infertility
Keywords: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vitamin D deficient patients: Serum 25-OH Vitamin D levels <20ng/L
- Vitamin D sufficient patients: Serum 25-OH Vitamin D levels ≥20ng/L

SUMMARY:
The role of vitamin D deficiency in female reproduction remains controversial. Early retrospective studies were inconsistent regarding the effect of serum 25-OH vitamin D levels on pregnancy rates in women undergoing in vitro fertilization (IVF), whereas two retrospective studies postulated that vitamin D deficiency may negatively affect pregnancy rates with an effect mediated through the endometrium.

Taking into account that knock-out experiments have shown that vitamin D receptor null mice not only experience uterine hypoplasia but also impaired folliculogenesis, it might be hypothesized that vitamin D deficiency may have a detrimental effect on female ovarian reserve. This may be further supported by previous reports demonstrating that serum 25-OH Vitamin D levels correlates with antimullerian hormone (AMH) levels in women of advanced reproductive age.

The aim of this study is to examine through a large set of prospectively recruited infertile women whether serum 25-OH-Vitamin D levels is related with the 2 most widely accepted biomarkers of ovarian reserve: serum AMH levels and antral follicle count (AFC).

ELIGIBILITY:
Inclusion Criteria:

infertile women less than 42 years old, undergoing their first treatment cycle in our institution

Exclusion Criteria:

vitamin D supplements, taking medication for systematic disease or having potential iatrogenic (e.g. ovarian surgery, gonadotoxic therapy) or known genetic cause of ovarian loss

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile women 18-43 years old undergoing IVF/ICSI
Sampling Method: Non-Probability Sample
Enrollment: 283 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Antimullerian hormone values in relation to vitamin D status | Between 0-28 days prior to having their 1st ultrasound scan for the determination of antral follicle count (AFC)
  On the day of the preliminary testing (irrespective of the day of the menstrual cycle) patients will have their serum 25-OH-vitamin D and antimullerian hormone levels determined. 25-OH-vitamin D and antimullerian hormone levels will be measured in samples retrieved on the same day
Antral follicle count in relation to vitamin D status | 2nd-3rd day of the menstrual cycle following the determination of vitamin D levels
  On the following cycle of the measurement of serum 25-OH-Vitamin D and AMH levels patient will have a transvaginal ultrasound to determine the antral follicle count (AFC)

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos P. Polyzos, MD PhD, Principal Investigator — Universitair Ziekenhuis Brussel; Arne Van de Vijver, MD, Principal Investigator — UZBrussel
Locations (1):
- Centre for Reproductive Medicine UZ Brussel, Brussels, Belgium

REFERENCES:
- [Background] Ozkan S, Jindal S, Greenseid K, Shu J, Zeitlian G, Hickmon C, Pal L. Replete vitamin D stores predict reproductive success following in vitro fertilization. Fertil Steril. 2010 Sep;94(4):1314-1319. doi: 10.1016/j.fertnstert.2009.05.019. Epub 2009 Jul 8. PMID 19589516
- [Background] Anifandis GM, Dafopoulos K, Messini CI, Chalvatzas N, Liakos N, Pournaras S, Messinis IE. Prognostic value of follicular fluid 25-OH vitamin D and glucose levels in the IVF outcome. Reprod Biol Endocrinol. 2010 Jul 28;8:91. doi: 10.1186/1477-7827-8-91. PMID 20667111
- [Background] Aleyasin A, Hosseini MA, Mahdavi A, Safdarian L, Fallahi P, Mohajeri MR, Abbasi M, Esfahani F. Predictive value of the level of vitamin D in follicular fluid on the outcome of assisted reproductive technology. Eur J Obstet Gynecol Reprod Biol. 2011 Nov;159(1):132-7. doi: 10.1016/j.ejogrb.2011.07.006. Epub 2011 Aug 10. PMID 21835540
- [Background] Rudick B, Ingles S, Chung K, Stanczyk F, Paulson R, Bendikson K. Characterizing the influence of vitamin D levels on IVF outcomes. Hum Reprod. 2012 Nov;27(11):3321-7. doi: 10.1093/humrep/des280. Epub 2012 Aug 21. PMID 22914766
- [Background] Rudick BJ, Ingles SA, Chung K, Stanczyk FZ, Paulson RJ, Bendikson KA. Influence of vitamin D levels on in vitro fertilization outcomes in donor-recipient cycles. Fertil Steril. 2014 Feb;101(2):447-52. doi: 10.1016/j.fertnstert.2013.10.008. Epub 2013 Nov 5. PMID 24210230
- [Background] Dennis NA, Houghton LA, Jones GT, van Rij AM, Morgan K, McLennan IS. The level of serum anti-Mullerian hormone correlates with vitamin D status in men and women but not in boys. J Clin Endocrinol Metab. 2012 Jul;97(7):2450-5. doi: 10.1210/jc.2012-1213. Epub 2012 Apr 16. PMID 22508713
- [Background] Merhi ZO, Seifer DB, Weedon J, Adeyemi O, Holman S, Anastos K, Golub ET, Young M, Karim R, Greenblatt R, Minkoff H. Circulating vitamin D correlates with serum antimullerian hormone levels in late-reproductive-aged women: Women's Interagency HIV Study. Fertil Steril. 2012 Jul;98(1):228-34. doi: 10.1016/j.fertnstert.2012.03.029. Epub 2012 Apr 10. PMID 22494925
- [Background] Yoshizawa T, Handa Y, Uematsu Y, Takeda S, Sekine K, Yoshihara Y, Kawakami T, Arioka K, Sato H, Uchiyama Y, Masushige S, Fukamizu A, Matsumoto T, Kato S. Mice lacking the vitamin D receptor exhibit impaired bone formation, uterine hypoplasia and growth retardation after weaning. Nat Genet. 1997 Aug;16(4):391-6. doi: 10.1038/ng0897-391. PMID 9241280